CLINICAL TRIAL: NCT04997551
Title: Double Blind Randomized Clinical Trial of Use of Colchicine Added to Standard Treatment in Hospitalized Patients With Covid-19 Infection
Brief Title: Double Blind Randomized Clinical Trial of Use of Colchicine Added to Standard Treatment in Hospitalized With Covid-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC CORONACOLCHI
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Infection
Keywords: covid-19; colchicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): EC Experimental group: colchicine for 2 weeks orally added to standard treatment.
  Interventions: Drug: Colchcine
- Placebo (Placebo Comparator): Control group: placebo for 2 weeks added to standard treatment.
  Interventions: Drug: Colchcine

INTERVENTIONS:
Drug: Colchcine — In patients not taking lopinavir / ritonavir or any other CYP3A4 or P-glycoprotein inhibitor drugs:
  * Day 1: 1 single dose of 1 mg orally, in a single dose.
  * Days 2 to 6: 0.5 mg every 12 hours v.o.
  * Days 7 to 14: 0.5 mg / 24 hours v.o. In patients taking drugs that inhibit the CYP3A4 system or the P-glycoprotein, these drugs will be attempted to be discontinued. The dose in these cases will be: o 0.5 mg every 72 hours v.o. while taking the drug that interacts.
  or 0.5 mg every 24 hours v.o. when, after suspending the interacting drug, at least 5 half-lives of the suspended drug have elapsed, from the last intake of said drug (in the case of lopinavir / ritonavir this would be a total of 24-30 hours) until the 14th day.
  In patients older than 80 years or patients with CKD-EPI estimated glomerular renal failure filtration rate between 30 and 50 ml / min / 1.73 m2), the colchicine / placebo dose will be:
  o Days 1 to 14: 0.5 mg / day

SUMMARY:
EC CORONACOLCHI is a multicenter, double-blind and randomized clinical trial with two branches. Patients who meet all the inclusion criteria and none of the exclusion criteria will be randomized 1: 1 to be included in one of the following groups:

* Experimental group: colchicine for 2 weeks orally at the doses described, added to the standard treatment of COVID-19.
* Control group: placebo for 2 weeks orally added to standard COVID-19 treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1 - Acute symptoms compatible with SARS-CoV-2 infection: fever, cough, myalgia, dysgeusia / ageusia, dyspnea, pulmonary infiltrates on X-ray / CT, or any sign / symptom attributable to said infection
* 2. Microbiologically confirmed infection by SARS-CoV-2 (PCR and / or CLIA or ELISA serology or with a valid microbiological diagnostic test with antigen test).
* 3.> 18 years.
* 4. <2 weeks from the onset of symptoms.
* 5. Admitted (with or without pneumonia) and ambulant (with pneumonia demonstrated by X-ray or CT)
* 6. Some analytical degree of moderate inflammation defined by PCR between 20 and 80 mg / L and / or ferritin between the high limit of normality (LAN) and 3 times said LAN
* 7. Signing of the Informed Consent, or acceptance of oral consent before witnesses.

Exclusion Criteria:

* 1. Drug allergy.
* 2. Intolerance to lactose and / or cow's milk proteins.
* 3. Renal failure with GFR <30 ml / min.
* 4. Liver cirrhosis or severe liver failure
* 5. Pregnancy or breastfeeding.
* 6. Blood dyscrasias or cardiac disorders that in the opinion of the investigator contraindicate the use of colchicine.
* 7. Pre-existing degenerative neuromuscular disease.
* 8. Acute or chronic diarrhea or malabsorptive syndrome that in the judgment of the clinician contraindicates the use of colchicine.
* 9. CRP> 80 mg / L or ferritin> 3 times LAN
* 10. Shock or hemodynamic instability.
* 11. Respiratory distress measured by PaO2 / FIO2 <300 or baseline O2 saturation ≤ 93%.
* 12. Patients undergoing mechanical ventilation.
* 13. Chronic treatment with any drug that, in the opinion of the investigator, interacts with colchicine and cannot be discontinued during the clinical trial, unacceptably increasing the risk of toxicity (digoxin, cyclosporine, etc.)
* 14. Have received any dose of colchicine, tocilizumab, any antiL6 or antiL1 drug.
* 15. Current treatment with corticosteroids (except chronic corticosteroid therapy without recent increase in dose).
* 16. Participation in any other clinical trial of patients with COVID-19.
* 17. Any other condition that, in the opinion of the investigator, contraindicates the use of colchicine or puts the subject at risk due to their participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who present death, need for mechanical ventilation or respiratory distress (Pa02 / FiO2 <300 or baseline O2 saturation ≤93%) on days +7, +14 and +30. | 30 days (from day +1 to day +30)
  Although the definition of respiratory distress usually includes a radiological criterion, as long as the oxygenation deficit is not attributable to another cause by the clinician, we do not consider it essential to perform a chest X-ray to confirm the diagnosis of distress because it does not correspond to clinical practice routine and the X-ray result does not change the patient's management.
Each of the items (proportion of patients who suffer death, need for mechanical ventilation and development of respiratory distress) separately on days +7, +14 and +30. | 30 days (from day +1 to day +30)

SECONDARY OUTCOMES:
Proportion of patients in each of the items of the clinical scale detailed below on days +3, +7, +14 and +30: | 30 days (from day +1 to day +30)
  1. Not hospitalized, usual activities not limited
  2. Not hospitalized with limitation for usual activities
  3. Hospitalized, without oxygen requirements
  4. Hospitalized with oxygen requirements
  5. Hospitalized with oxygen in a reservoir, non-invasive mechanical ventilation or high-flow oxygen device
  6. Hospitalized with the need for invasive mechanical ventilation
  7. Deceased
Time (days) until death | 30 days (from day +1 to day +30)
Proportion of patients in whom fever ≥37.8 ºC persists on days +3, +7, +14 and +30. | 30 days (from day +1 to day +30)
Evolution of the levels of C-Reactive Protein (CRP), LDH, D-dimer, ferritin, lymphocytes on days +3, +7, +14 and +30. | 30 days (from day +1 to day +30)
Proportion of patients who have received tocilizumab / other antiL6 or antiL1 drug / corticosteroids on days +3, +7, +14 and +30. | 30 days (from day +1 to day +30)
Proportion of patients experiencing serious unexpected adverse reactions that require discontinuation of the investigational product. | 30 days (from day +1 to day +30)

CONTACTS AND LOCATIONS:
Locations (1):
- Biodonostia Health Research Institute, San Sebastián, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: No